CLINICAL TRIAL: NCT03568175
Title: A Phase II/III Study of JR-141 in Patients With Mucopolysaccharidosis II
Brief Title: A Study of JR-141 in Patients With Mucopolysaccharidosis II
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JR-141-301
Record Dates: First submitted 2018-06-01; First posted 2018-06-26 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Mucopolysaccharidosis II
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JR-141 2.0 mg/kg/week (Experimental)
  Interventions: Drug: JR-141

INTERVENTIONS:
Drug: JR-141 — IV infusion, 2.0 mg/kg/week

SUMMARY:
A Phase II/ III multicenter, open-label, single-group, designed to evaluate the efficacy and safety of study drug for the treatment of the MPS II.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of providing written consent by himself (not mandatory for those aged under 20 years at the time of informed consent process, or those who is impossible to obtain consent from the patient himself due to intellectual disabilities associated with MPS II.)
2. In the case of a patient who is under the age of 20 years or from whom it is not possible to obtain consent due to intellectual disabilities associated with MPS II, he may be included if written consent can be provided by legal representative (however, written consent should be obtained from the patient himself too, whenever possible)
3. Males with confirmed diagnosis of MPS II, based on deficient activity of iduronate-2-sulfatase (IDS) in leucocytes, plasma or fibroblasts and/or pathogenic mutations identified in the IDS gene, etc.
4. Naïve patients or patients who are receiving stable enzyme replacement therapy with Elaprase for more than 8 weeks before the observational period starts.

Exclusion Criteria:

1. Previous engrafted HSCT, excluding those who need enzyme replacement therapy even after HSCT.
2. Judged by the investigator or subinvestigator as being unable to undergo lumbar puncture, including those who have difficulties in taking position for lumbar puncture due to joint contracture or those who are likely experience difficulty breathing during the lumbar puncture process.
3. Judged by the investigator or subinvestigator to be ineligible to participate in the study due to a history of serious drug allergy or sensitivity.
4. Patients who have received other investigational product within 4 months before enrollment in the study.
5. Otherwise judged by the investigator or subinvestigator to be ineligible to participate in the study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Heparan Sulfate Levels in Cerebrospinal Fluid | Baseline to 52 weeks

SECONDARY OUTCOMES:
Change From Baseline in Serum Heparan Sulfate Levels. | Baseline, 24-26 weeks, 50-52 weeks
Change From Baseline in Serum Dermatan Sulfate Levels. | Baseline, 24-26 weeks, 50-52 weeks
Change From Baseline in Urinary Heparan Sulfate Levels. | Baseline, 25 weeks, 52 weeks
Change From Baseline in Urinary Dermatan Sulfate Levels. | Baseline, 25 weeks, 52 weeks
Change From Baseline in Liver Volumes. | Baseline, 25 weeks, 52 weeks
Change From Baseline in Spleen Volumes. | Baseline, 25 weeks, 52 weeks
Change From Baseline in Cardiac Function. | Baseline, 25 weeks, 52 weeks
Change From Baseline in 6-minute Walk Test Distance. | Baseline, 25 weeks, 52 weeks
  Item 9 will be administrated only in patients judged by the investigator or subinvestigator to be possible to perform the 6-minutes walk test
Change From Baseline in Joint Range of Motion. | Baseline, 25 weeks, 52 weeks
Change From Baseline in Heparan Sulfate Levels in Cerebrospinal Fluid. | Baseline to 25 weeks
Change From Baseline in Dermatan Sulfate Levels in Cerebrospinal Fluid. | Baseline, 25 weeks, 52 weeks
Change from Baseline in Neurocognitive Testing (Kyoto Scale of Psychological Development 2001) | 25, 52 weeks
Change from Baseline in Adaptive Behavioral Testing ( Vineland Adaptive Behavior Scales Second Edition. ) | 25, 52 weeks
Drug concentration in Cerebrospinal Fluid. | 25, 52*weeks
  *Drug concentration in Cerebrospinal Fluid at 52 Weeks is applicable only for subjects to be enrolled in extension study .

CONTACTS AND LOCATIONS:
Locations (19):
- Japan (19):
  - Fukui Clinical site, Fukui
  - Fukuoka Clinical site 2, Fukuoka
  - Fukuoka Clinical site, Fukuoka
  - Gifu Clinical site, Gifu
  - Hokkaido Clinical site, Hokkaido
  - Kanagawa Clinical site, Kanagawa
  - Kumamoto Clinical site, Kumamoto
  - Okayama Clinical site, Okayama
  - Okayama Clinical site 2, Okayama
  - Okinawa Clinical site, Okinawa
  - Osaka Clinical site 3, Osaka
  - Osaka Clinical site 2, Osaka
  - Osaka Clinical site, Osaka
  - Saitama Clinical site, Saitama
  - Shizuoka Clinical site, Shizuoka
  - Shizuoka Clinical site 2, Shizuoka
  - Tochigi Clinical site, Tochigi
  - Tokyo Clinical site, Tokyo
  - Tottori Clinical site, Tottori

REFERENCES:
- See also: A Phase 2/3 Trial of Pabinafusp Alfa, IDS Fused with Anti-Human Transferrin Receptor Antibody, Targeting Neurodegeneration in MPS-II — https://pubmed.ncbi.nlm.nih.gov/33038326/